CLINICAL TRIAL: NCT01366014
Title: A Study of ARRY-371797 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARRAY-797-223; C4411007 (Other: Pfizer)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; pain; NSAID
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — ARRY-371797; Oxycodone; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARRY-371797 (Experimental)
  Interventions: Drug: ARRY-371797, p38 inhibitor; oral
- Oxycodone HCl ER (Active Comparator)
  Interventions: Drug: Oxycodone hydrochloride (HCl) extended release (ER), opioid agonist; oral
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; oral

INTERVENTIONS:
Drug: ARRY-371797, p38 inhibitor; oral — multiple dose, single schedule
  Arms: ARRY-371797
Drug: Oxycodone hydrochloride (HCl) extended release (ER), opioid agonist; oral — multiple dose, single schedule
  Arms: Oxycodone HCl ER
Drug: Placebo; oral — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2 study, involving a 4-week treatment period, designed to test the ability of investigational study drug ARRY-371797 to reduce pain in patients with moderate to severe pain due to osteoarthritis (OA) of the knee, and to further evaluate the drug's safety. Approximately 150 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of OA of the knee, based on American College of Rheumatology (ACR) criteria, confirmed by X-ray (K-L Grade II/III within the last year).
* At least moderate or severe pain due to OA in one knee.
* On nonsteroidal anti-inflammatory drug (NSAID) 28 days previous to study start and willing to continue on NSAID throughout study.
* Discontinuation of opioids prior to study start.
* Additional criteria exist.

Key Exclusion Criteria:

* Current or recent infection in the last 7 days; infection requiring hospitalization or parenteral antibiotics within the last 6 months; history of or currently active tuberculosis, hepatitis B or C, or human immunodeficiency virus (HIV).
* Surgery on the index knee within the previous 6 months.
* Trauma or other surgeries within the previous 8 weeks.
* Specific abnormal laboratory values or electrocardiogram abnormalities.
* Gastrointestinal surgery that may interfere with motility or absorption.
* On non-stable dose of bisphosphonates, or any prior denosumab or parathyroid hormone (PTH) therapies.
* Prior parenteral tumor necrosis factor (TNF) inhibitor or anti-nerve growth factor (NGF) therapies.
* Intramuscular, intravenous or oral corticosteroids within the previous 6 weeks.
* Intra-articular corticosteroids in the index knee within the previous 8 weeks or viscosupplementation in the index knee within the previous 4 months.
* Currently enrolled in or participated in another clinical trial within the previous 3 months.
* Additional criteria exist.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the study drug (versus placebo) in terms of change from baseline to week 4 in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score (index knee). | 4 weeks

SECONDARY OUTCOMES:
Assess the efficacy of the study drug (versus placebo) in terms of change from baseline to week 4 in the WOMAC stiffness and physical function subscale scores (index knee). | 4 weeks
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, electrocardiograms and vital signs. | 5 weeks
Characterize the pharmacokinetics of the study drug and metabolite as determined by plasma concentrations. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Kenosha, Wisconsin